# Examining Patient Involvement Patterns and Trends in Participation in Bone Cancer Clinical Trials

This is an Informed Consent Form For Bone Cancer Patients in <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: September 30, 2023

Recognizing the Significance of This Informed Consent Form

If you are tasked with filling out this paperwork, it indicates your potential eligibility for participation in a unique observational clinical study aimed at bone cancer patients. This in-depth guide elucidates the study's core objectives, detailed execution strategy, and various consequences, both favorable and potentially adverse. Prior to making a decision, it is imperative to thoroughly explore the details of your potential participation, and seeking advice from a reliable source can offer valuable perspectives. Should any portion of this document seem unclear or if questions arise, rest assured that the researcher is accessible to provide clarification.

The Significance of Clinical Trials in the Context of Bone Cancer

Bone cancer is a rare type of cancer that begins in the bone tissue. It can develop in any bone in the body but most commonly affects the long bones of the arms and legs. There are several types of bone cancer, with the most common being osteosarcoma and chondrosarcoma.

The exact cause of bone cancer is often unknown, but some genetic and environmental factors may play a role. Treatment for bone cancer typically involves a combination of surgery, radiation therapy, and chemotherapy, depending on the type and stage of cancer. Prognosis varies depending on factors such as the type of bone cancer, its

stage at diagnosis, and the patient's overall health. Early detection and prompt treatment can improve outcomes for individuals with bone cancer.

Clinical studies, with a distinct focus on bone cancer, play a crucial role in evaluating the safety and effectiveness of novel treatments for this disease. These trials serve as instrumental means to determine whether new medications surpass conventional therapies, providing substantial evidence for their broader adoption.

What sets this particular study apart is its central emphasis on the firsthand experiences of individuals grappling with bone cancer, actively participating in a clinical trial featuring medicinal interventions. The primary objective is to meticulously scrutinize trial completion rates and voluntary withdrawals within this specific patient group.

### Exploring the Core of Observational Trials

Venturing into this medical trial involves immersing oneself in an observational study, a unique facet of clinical research meticulously tailored to unveil insights through unobtrusive observation of patients while preserving their treatment regimens.

Researchers will exclusively observe your journey, carefully assessing the outcomes of your condition without any interventions. This specific trial design holds paramount importance in deepening our understanding of the inherent progression of a particular medical ailment and its consequences for individuals affected by it. By actively participating in this observational study, you assume a pivotal role in expanding the frontiers of medical knowledge and driving advancements in the care provided to those enduring the same condition.

# Setting This Trial Apart from Other Bone Cancer Clinical Investigations

Recognizing the distinctive aspects of this research study is of utmost importance. It operates solely on an observational basis, indicating that your participation will not involve any specific treatments or interventions. To arrive at an informed decision regarding potential involvement in a clinical trial, it is essential to comprehend the spectrum of bone cancer clinical investigations, including interventional studies in which participants undergo diverse treatment regimens.

Making an informed choice concerning your potential participation in a clinical trial requires an active approach that includes research and a comparison of various trials.

Resources like Clinicaltrials.gov and similar platforms offer a wealth of information on research pertaining to bone cancer. Moreover, Power's specialized web platform provides a comprehensive list of ongoing bone cancer clinical trials actively recruiting volunteers. Arming yourself with thorough research and a comprehensive understanding of different clinical trial categories empowers you to decisively shape your participation decision.

### Active Participation in Clinical Trial Surveys: Your Choice

We warmly invite you to actively share your experiences as a vital part of this observational clinical investigation. This endeavor involves completing questionnaires every two weeks, taking approximately 20-30 minutes of your valuable time. Furthermore, we are fully equipped to conduct check-in calls at quarterly intervals, a practice that will continue throughout your participation in the trial.

It is essential to emphasize that your involvement in the survey phase of the trial is entirely at your discretion. You have the autonomy to decide whether to respond to specific questions or complete the entire questionnaire. Additionally, you maintain the freedom to withdraw from the trial at any time, should you choose to do so. Recognizing that the decision to participate in a clinical study is a deeply personal one, we are committed to providing the necessary support. Your privacy and comfort are of the utmost importance to us, and we are dedicated to respecting and assisting your decision-making process throughout the trial.

# Preserving the Privacy of Your Responses

Preserving the full confidentiality of your information is of utmost importance during the course of this research study. To protect your anonymity, we respectfully request that you refrain from including any personal or identifiable details in your questionnaire responses. The dedicated research team is unwavering in their dedication to enhancing the protection of your privacy. However, it's essential to recognize that specific legal scenarios may arise, necessitating the sharing of personal data.

Acknowledging Possible Health Implications

Despite the substantial strides made by clinical trials, it is crucial to acknowledge the possible health implications that participants may encounter, particularly in studies assessing new medications.

Nonetheless, our approach in observational clinical research takes a distinct route, deliberately mitigating these implications by refraining from the application of experimental therapies to participants. Our primary priority is rigorous monitoring and outcome evaluation, ensuring the avoidance of any undue health risks.

#### Foreseeing Possible Advantages

Though immediate advantages may not be readily discernible for participants in this observational clinical research, their participation holds the potential to exert a substantial impact on others. The information collected from participants will be leveraged to enhance future approaches to recruiting individuals with bone cancer, potentially widening the scope of medical exploration. Those who undertake this therapeutic expedition have the ability to spark substantial transformations in the landscape of medical research, potentially charting the course for future bone cancer patients.

# Fostering Inclusivity in Clinical Trials

Numerous online avenues eagerly invite your active participation if you are motivated by an unquenchable curiosity to delve into the intricate subject of diversity within clinical trials.

Whether your goal is to gain insight into the intricacies of the challenges and opportunities linked to clinical trial diversity or to broaden your own perspectives, the following resources could prove immensely beneficial:

Patel, Vimla L., José F. Arocha, Melissa Diermeier, Jacques How, and Christel Mottur-Pilson. "Cognitive psychological studies of representation and use of clinical practice guidelines." *International Journal of Medical Informatics* 63, no. 3 (2001): 147-167.

<u>Bibbins-Domingo, Kirsten, and Alex Helman. "Improving representation in clinical trials and research: building research equity for women and underrepresented groups."</u>
(2022).

#### Validation of Informed Consent

I hereby validate that I have dedicated sufficient time to grasp and internalize the information outlined in the informed consent form. This comprehension has been achieved through either independent review or with the guidance of a trusted individual who has elucidated its contents to me. All of my questions and concerns have been meticulously addressed to my utmost satisfaction.

I am fully conscious that my participation in this study is a result of my own volition, and I retain the sole authority to withdraw my consent without any obligation to provide reasons or assume financial responsibilities. I have received assurance that a copy of this informed consent form will be provided to me for my personal records.

After careful deliberation and a comprehensive review of all the materials presented to me, I hereby grant my consent to participate in this study, signifying my informed and autonomous decision.

| Participant Name |
|-----------------------|
| Participant Signature |
| Date |

Confirmation by Informed Consent Facilitator

I confirm that I have engaged in a comprehensive discussion with the participant, meticulously elucidating the intricacies encompassed within this written document. My objective was to ensure that the participant possessed a thorough understanding of the

primary research goals, the methodology employed, potential risks and benefits, and other essential components inherent to the bone cancer clinical trial.

The participant was afforded ample opportunity to pose questions and express concerns or seek clarifications. It is imperative to underscore that the participant's involvement in this study is entirely voluntary, and they retain the unimpeded right to withdraw at any time, for any reason, without incurring any financial obligations.

Following the participant's granting of consent, a diligently maintained duplicate of this written document was provided to them, serving as a repository for their specific information.

| Printed Name of Assisting Researcher |
|--------------------------------------|
| Signature of Assisting Researcher |
| Date |